CLINICAL TRIAL: NCT01031888
Title: Phase 1 Study of Topical Autologous Insulin Application for the Treatment of Corneal Epithelium Defect After Ocular Surgeries
Brief Title: Topical Autologous Insulin Application for the Treatment of Corneal Epithelium Defect After Ocular Surgeries
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Wei-Li Chen/Assistant Professor, National Taiwan University, Department of Ophthalmology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 200803017M
Record Dates: First submitted 2009-12-14; First posted 2009-12-15 (Estimated); Last update posted 2009-12-15 (Estimated); Status verified 2009-12

CONDITIONS: Corneal Epithelial Defects After Ocular Surgeries
Keywords: Corneal re-epithelialization; Topical insulin application; pars planar vitrectomy; diabetic retinopathy; penetrating keratoplasty
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator): Corneal epithelial wound healing in patients who received pars planar vitrectomy (PPV) for diabetic retinopathy receiving topical insulin eye drops in addition to conventional postoperative eye drops
  Interventions: Drug: Topical insulin eye drops
- 2 (Active Comparator): Corneal epithelial wound healing in patients who received pars planar vitrectomy (PPV) for penetrating keratoplasty receiving topical insulin eye drops in addition to conventional postoperative eye drops
  Interventions: Drug: Topical insulin eye drops
- 3 (Placebo Comparator): Corneal epithelial wound healing in patients who received pars planar vitrectomy (PPV) for diabetic retinopathy treated with conventional postoperative eye drops
  Interventions: Drug: Conventional postoperative eye drops
- 4 (Placebo Comparator): corneal epithelial wound healing in patients who received pars planar vitrectomy (PPV) for penetrating keratoplasty receiving conventional postoperative eye drops
  Interventions: Drug: Conventional postoperative eye drops

INTERVENTIONS:
Drug: Topical insulin eye drops — Regular insulin injection diluted to 100U/ml After the day of surgery, besides topical steroid, antibiotic and mydriatics, the patient receives topical insulin eye drops every two hours, except from 10pm to 8am, until the epithelial defect is totally closed
  Arms: 1; 2
Drug: Conventional postoperative eye drops — topical steroid, antibiotic and mydriatics
  Arms: 3; 4

SUMMARY:
Topical insulin application has been proved recently to increase corneal reepithelization rate over diabetic animals. However, its effectiveness on corneal epithelial wound healing in patients who received pars planar vitrectomy (PPV) for diabetic retinopathy and penetrating keratoplasty has not been reported. In this study, we plan to perform a prospective randomized study to determine the effectiveness of topical insulin as a primary treatment for corneal epithelial defect in patients undergoing vitrectomy for diabetic retinopathy and penetrating keratoplasty. All patients enrolled in this study have received corneal epithelial debridement at the end of the ocular surgeries, namely PPV for diabetic retinopathy and penetrating keratoplasty. The patients were randomized into two treatment groups. In the control group, the patients receive conventional postoperative eye drops including topical steroid, antibiotic and mydriatics. In the experimental group, the patients receive topical insulin eye drops in addition to conventional postoperative eye drops. The duration for the corneal surface to completely re-epithelize, the incidence of corneal complications due to delayed surface re-epithelization (e.g. infectious corneal ulcer, corneal melting, sterile corneal ulcer, corneal neovascularization), and the incidence of recurrent epithelial break down after initial epithelization will be compared between these two groups. Patients undergoing PPV for diabetic retinopathy and penetrating keratoplasty will be compared separately.

DETAILED DESCRIPTION:
Purpose: To evaluate the treatment effects of topical insulin eye drops for promoting corneal epithelium wound healing in patients receiving pars planar vitrectomy (PPV) for diabetic retinopathy and penetrating keratoplasty.

Background: During PPV for diabetic retinopathy retinopathy and penetrating keratoplasty, removal of the edematous corneal epithelial layer was usually required in order to obtain a better surgical view1 or enhance the postoperative epithelial wound healing process. However, delayed epithelial healing was frequently found in these patients after surgeries. In addition, corneal epithelial defect is also frequent found in diabetic patients after PPV even corneal epithelial debridement is not performed during the operation. Topical insulin application has been known to increase corneal reepithelization rate over diabetic animals, has is known to have no influence on systemic glucose level in humans and animals. In this study, we plan to perform a prospective randomized study to determine the effectiveness of topical insulin eye drops as a primary treatment in corneal epithelial defect following vitrectomy in diabetic patients and penetrating keratoplasty.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients with proliferative retinopathy receiving PPV
* Patients qualified for penetrating keratoplasty
* DM control blood sugar AC < 200mg/dl
* no limbus defect
* no glaucoma before and after surgery
* Patients willing to receive surgery, blood drawl and OPD follow up
* no previous corneal epithelial defect or disease

Exclusion Criteria:

* Limbus defect
* postsurgical use of other eye drops
* incomplete eyelid closure
* glaucoma
* unable to be followed up postoperatively
* poor visual acuity or poor prognostic visual acuity
* corneoneuropathy
* severe dry eye syndrome
* pregnant
* receive eye surgery within one month after the previous eye surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-03; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Duration for the corneal surface to completely re-epithelize | 1week, 2 weeks, 1 month, 2 month, 3 month, 6 month

SECONDARY OUTCOMES:
Incidence of corneal complications due to delayed surface re-epithelization (e.g. infectious corneal ulcer, corneal melting, sterile corneal ulcer, corneal neovascularization) | 1 week, 2 weeks, 1 month, 2 month, 3 month, 6 month
Incidence of recurrent epithelial break down after initial epithelization | 1 week, 2 weeks, 1 month, 2 month, 3 month, 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Li Chen, MD, PhD, Principal Investigator — National Taiwan University Hospital, department of Ophthalmology
Locations (1):
- National Taiwan University Hospital, department of Ophthalmology, Taipei, Taiwan